CLINICAL TRIAL: NCT00456625
Title: To Evaluate Immune Response to a Hepatitis B Vaccine (Engerix™-B ) Challenge Dose in Healthy Subjects Who Received GSK Biologicals' Hepatitis B Vaccine (Engerix™-B ) Approximately 20 Years Ago as Primary Vaccination at 0, 1, 2 and 12 Months.
Brief Title: Immune Response to Hepatitis B Vaccine Challenge Dose in Subjects Who Received a Primary Neonatal Hepatitis B Vaccine.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 108984
Record Dates: First submitted 2007-04-04; First posted 2007-04-05 (Estimated); Results first posted 2009-05-15 (Estimated); Last update posted 2016-12-16 (Estimated); Status verified 2016-11

CONDITIONS: Hepatitis B
Keywords: Hepatitis B vaccine; Challenge dose
MeSH Terms: conditions — Hepatitis B | interventions — Hepatitis B Vaccines

ARMS (1):
- Group Engerix™-B (Experimental): Subjects received a dose of Hepatitis B vaccine approximately 20 years after the primary neonatal vaccination
  Interventions: Biological: Engerix™-B

INTERVENTIONS:
Biological: Engerix™-B — Intramuscular injection, 1 dose
  Other Names: Hepatitis B vaccine

SUMMARY:
The current study will evaluate immunological memory to hepatitis B antigen in subjects who received primary neonatal vaccination of hepatitis B vaccine (Engerix™-B ), 20 years ago in the primary study and who have anti-HBs antibody concentrations < pre-defined cut-off values at the previous long-term time point. All participating subjects will receive a challenge dose of hepatitis B vaccine. Subjects will be aged approximately 20-21 years at the time of this study. No new subjects will be recruited in this long-term follow-up study. Blood sampling will be done one month after the administration of the challenge dose. The Protocol Posting has been updated in order to comply with the FDA Amendment Act, Sep 2007.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes that they can and will comply with the requirements of the protocol should be enrolled in the study.
* A male or female adult who received the complete neonatal primary vaccination course of hepatitis B vaccine in primary study approximately 20 years earlier.
* Documented level of anti-HBs antibody concentrations < specified concentration at the previous long-term time point for which serological results are available for that subject.
* Written informed consent obtained from the subject.
* Healthy subjects as established by medical history and clinical examination before entering into the study.
* If the subject is female, she must be of non-childbearing potential or if she is of childbearing potential, she must practice adequate contraception for 30 days prior to vaccination, have a negative pregnancy test and continue such precautions for 2 months after completion of the hepatitis B challenge dose.

Exclusion Criteria:

* Chronic administration (defined as more than 14 days) of immunosuppressants or other immune-modifying drugs within six months prior to the hepatitis B vaccine challenge dose.
* Administration of a vaccine not foreseen by the study protocol during the study period.
* Administration of immunoglobulins and/or any blood products during the study period.
* Drug and/or alcohol abuse.

Ages: 20 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 76 (Actual)
Dates: Start 2007-04; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Poovorawan Y, Chongsrisawat V, Theamboonlers A, Bock HL, Leyssen M, Jacquet JM. Persistence of antibodies and immune memory to hepatitis B vaccine 20 years after infant vaccination in Thailand. Vaccine. 2010 Jan 8;28(3):730-6. doi: 10.1016/j.vaccine.2009.10.074. Epub 2009 Nov 3. PMID 19892043
- [Background] Poovorawan Y, Chongsrisawat V, Theamboonlers A, Leroux-Roels G, Kuriyakose S, Leyssen M, Jacquet JM. Evidence of protection against clinical and chronic hepatitis B infection 20 years after infant vaccination in a high endemicity region. J Viral Hepat. 2011 May;18(5):369-75. doi: 10.1111/j.1365-2893.2010.01312.x. PMID 20384962
- [Background] Poovorawan Y et al. 20-year follow-up of immunogenicity and efficacy of infant hepatitis B vaccination. Abstract presented at the 6th World Congress of the World Society for Pediatric Infectious Diseases (WSPID). Buenos Aires, Argentina, 18-22 November 2009.
- [Background] Poovorawan Y et al. 20-year persistence of immune response to infant hepatitis B vaccination in a high endemicity region. Abstract presented at the 13th International Symposium on Viral Hepatitis and Liver Disease (ISVHLD), Washington DC, US, 20-24 March 2009.
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Informed Consent Form: 108984 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 108984 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 108984 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 108984 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 108984 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 108984 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 108984 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Group Engerix™-B
Started | 76
Completed | 76
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Group Engerix™-B
Number analyzed (Participants) | 76
Age, Continuous [Mean (Standard Deviation); unit: years] | 19.9 (0.59)
Gender [Count of Participants; unit: Participants]
  Female | 36
  Male | 40

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Anti-hepatitis B Surface Antigen (Anti-HBs) Antibody Concentrations Above Specific Cut-off Values
Description: The cut-off values assessed include: ≥ 3.3 Milli International Units per Milliliter (mIU/mL), ≥ 10 mIU/mL, and ≥ 100 mIU/mL.
Time Frame: One month after the hepatitis B vaccine challenge dose
Population: The analysis was performed on the According-to-Protocol (ATP) cohort for immunogenicity (including all evaluable subjects who had received the challenge dose of hepatitis B vaccine and for whom immunogenicity data were available at the post-hepatitis B vaccine challenge dose timepoint).
Measure: Number; unit: participants
Arm/Group | Group Engerix™-B
Number analyzed (Participants) | 72
participants
  ≥ 3.3 mIU/mL | 72
  ≥ 10 mIU/mL | 71
  ≥ 100 mIU/mL | 64

2. Secondary Outcome: Occurrence, Intensity and Relationship to Vaccination of Unsolicited Adverse Events (AEs)
Description: An AE is any untoward medical occurrence in a clinical investigation subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.
  An AE is considered severe if it prevents normal, everyday activities.
Time Frame: During the 31-day follow-up period after the challenge dose of hepatitis B vaccine.
Measure: Number; unit: participants
Arm/Group | Group Engerix™-B
Number analyzed (Participants) | 76
participants
  Any AEs | 1
  Severe AEs | 0
  Related AEs | 0

3. Secondary Outcome: Number of Participants Reporting Any Serious Adverse Events (SAEs).
Description: An SAE is any untoward medical occurrence that:
  results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect in the offspring of a study subject, or may evolve into one of the outcomes listed above.
Time Frame: Up to 1 month after the challenge dose.
Measure: Number; unit: participants
Arm/Group | Group Engerix™-B
Number analyzed (Participants) | 76
participants | 0

ADVERSE EVENTS:
Arm/Group | Group Engerix™-B
Serious Adverse Events (participants affected / at risk) | 0/76
Other Adverse Events (participants affected / at risk) | 0/76

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.